CLINICAL TRIAL: NCT04823975
Title: Improving Health Insurance Literacy Among Utah's Hispanic Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Anne Kirchhoff, Associate Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB_00138483; UL1TR002538 (NIH)
Record Dates: First submitted 2021-03-19; First posted 2021-04-01 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: Health Insurance; Literacy
MeSH Terms: conditions — Behavior; Literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIEP intervention (Experimental): Participants will be given the health insurance intervention from Utah Health Policy Project staff, a 60 minute long, educational learning session.
  Interventions: Behavioral: Health Insurance Education Program (HIEP)

INTERVENTIONS:
Behavioral: Health Insurance Education Program (HIEP) — [See arm/group description]

SUMMARY:
This is a test of an existing health insurance education program (HIEP) in the Utah Hispanic community (aged 18-64). The study will evaluate whether the HIEP delivered by Utah Health Policy Project (UHPP) staff improves participants' health insurance and cost-related literacy. Participants will complete a brief baseline survey, be guided through the HIEP by UHPP staff, and complete a brief survey after completing the sessions.

DETAILED DESCRIPTION:
The goal of this research is to refine and pilot test an existing health insurance education program (HIEP) to improve health insurance and cost-related literacy among the Hispanic community in Utah. This study will be conducted in conjunction with the Utah Health Policy Project, which has long been active in the Hispanic community and has been instrumental in reducing the number of uninsured adults and children in Utah. Initially, community and key-informant feedback on how to best adapt this intervention to the Hispanic community, including what topics are most important, and how the intervention should be delivered, will be obtained. After the HIEP is adapted accordingly, it will be investigated to see if it improves participants' health insurance and cost-related literacy.

Upon enrollment, participants will fill out a survey containing questions about their current health insurance, employment, demographics, acculturation, preferred language and health insurance knowledge. Participants will then receive an educational session surrounding health insurance use and laws. This educational sessions will be conducted, in person, over video conference calls, or over the telephone, and will cover:

* Overview of health insurance options and understanding of insurance and costs
* Learning about types of insurance coverage and how to select/access coverage
* Navigating one's coverage plan
* Managing care costs

This sessions will be 60 minutes.

After completing the HIEP participants will be given a second survey including similar questions to those in the first survey. This survey will include questions to obtain feedback on the acceptability of the content and potential implementation issue areas, as well as any discordance in cultural values, beliefs, or feelings about health insurance.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Hispanic
* Resident of Utah
* Primary Policy Holder
* Recently enrolled in health insurance within the past year

Exclusion Criteria:

* Younger than 18 years of age
* Not Hispanic or Latino/Latina in origin
* Non-Utah resident
* Non Policy holder
* Not recently enrolled in health insurance

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne C Kirchhoff, PhD, Principal Investigator — University of Utah Department of Pediatrics
Locations (1):
- Utah Health Policy Project, West Valley City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- HIEP Intervention: Participants will be given the health insurance intervention from Utah Health Policy Project staff, which includes a, 60 minute long, educational learning session.
  Health Insurance Education Program (HIEP): [See arm/group description]
Period: Overall Study
Arm/Group | HIEP Intervention
Started | 12
Completed | 9
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | HIEP Intervention
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants] — Population: Two participants did not provide the study with their age.
  Participants
    number analyzed (Participants) | 10
    <=18 years | 0
    Between 18 and 65 years | 10
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Two participants did not provide the study with their age.
  years
    number analyzed (Participants) | 10
    (all) | 35.4 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Health Insurance Literacy Measure (Limited number of items) [Mean (Standard Deviation); unit: units on a scale] — Limited number of item from the Health Insurance Literacy Measure. Higher score are better; scores could range from 6 to 24
  units on a scale | 14.67 (5.65)

OUTCOME MEASURES:

1. Primary Outcome: Number of Enrolled Individuals
Description: A count of the individuals who enrolled in the study.
Time Frame: Post-Assessment survey (Weeks 19 (+/- 2 weeks))
Measure: Number; unit: participants
Arm/Group | HIEP Intervention
Number analyzed (Participants) | 12
participants | 9

2. Primary Outcome: Number of Completed Sessions Per Enrolled Individual
Description: The average number of completed sessions per individual enrolled in the study.
Time Frame: Post-Assessment survey (Weeks 19 (+/- 2 weeks))
Measure: Mean (Standard Deviation); unit: Education sessions completed
Arm/Group | HIEP Intervention
Number analyzed (Participants) | 12
Education sessions completed | 0.83 (0.39)

3. Secondary Outcome: Changes in the Health Insurance Literacy Measure Based on Age Group
Description: Differences between Health Insurance Literacy Measure (HILM) reported at the baseline and post-assessment survey. Differences will be examined by age. Lower scores indicate lower health insurance literacy, higher scores are better. Scores could range from 6 to 24. We report on a limited number of item from the Health Insurance Literacy Measure. We will report mean and standard deviation at both time points.
Time Frame: Baseline (Week 0) and Post Assessment survey (Weeks 19 (+/- 2 weeks))
Population: Analysis was run on individuals who completed both the baseline and the followup survey and who reported their age.
Measure: Mean (Standard Deviation); unit: Change in score on a scale
Groups:
- HIEP Intervention: Participants will be given the health insurance intervention from Utah Health Policy Project staff, which includes one, 30 minute long, educational learning session.
  Health Insurance Education Program (HIEP): [See arm/group description]
Arm/Group | HIEP Intervention
Number analyzed (Participants) | 8
Change in score on a scale
  Age 18-25: number analyzed (Participants) | 2
  Age 18-25 | 10.5 (6.36)
  Age 26-64: number analyzed (Participants) | 6
  Age 26-64 | 4.33 (3.50)

4. Secondary Outcome: Changes in the Health Insurance Literacy Measure Based on Language Spoken
Description: Differences between Health Insurance Literacy Measure (HILM) reported at the baseline and post-assessment survey. Differences will be examined by language spoken. Lower scores indicate lower health insurance literacy, higher scores are better. Scores could range from 6 to 24. We report on a limited number of item from the Health Insurance Literacy Measure. We will report mean and standard deviation at both time points.
Time Frame: Baseline (Week 0) and Post Assessment survey (Weeks 19 (+/- 2 weeks))
Population: Analysis was completed for individuals who completed both the baseline and the followup survey.
Measure: Mean (Standard Deviation); unit: Change in score on a scale
Arm/Group | HIEP Intervention
Number analyzed (Participants) | 9
Change in score on a scale
  English Speaking Preferred: number analyzed (Participants) | 5
  English Speaking Preferred | 9.00 (4.06)
  Spanish Speaking Preferred: number analyzed (Participants) | 4
  Spanish Speaking Preferred | 3.25 (3.77)

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored for this study.
Description: As this study was an educational intervention on health insurance, mortality, serious and non-serious adverse events were not monitored/assessed.
Arm/Group | HIEP Intervention
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT04823975/Prot_SAP_002.pdf
  • Informed Consent Form (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT04823975/ICF_001.pdf